CLINICAL TRIAL: NCT03792243
Title: Outcomes After Parastomal Hernia Repair
Status: Completed | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: Danish Hernia Database (Unknown)
Responsible Party: Principal Investigator, Frederik Helgstrand, MD, DMSc, Ass prof, Zealand University Hospital
Other Study IDs: Parastomalhernia 2019
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Parastomal Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parastomal hernia: Patients undergoing parastomal hernia repair in Denmark between 2007 and 2017
  Interventions: Procedure: Complication

INTERVENTIONS:
Procedure: Complication — Readmission, reoperation

SUMMARY:
The aim of the current study is to evaluate the overall outcomes after parastomal hernia repairs in Denmark from 2007-2017 using data from the Danish Hernia Database and Danish Patients Registry. Specifically, the readmission and reoperation rates will be evaluated.

DETAILED DESCRIPTION:
The Danish Hernia Database covers about 80% of all ventral hernia repairs performed in Denmark. Data on size of hernia, type of surgery, type of mesh and fixation method is available from the Danish Hernia Database. All healthcare services in Denmark are registered in the Danish National Patients Registry and data on 30-day readmission rate, readmission diagnosis and reoperation is found here. Each Danish citizen has a unique personal identification number and by merging data from the Danish Hernia Database and National Patients Registry, nationwide data on parastomal hernia repairs is available. The aim of the current study is to evaluate the overall outcomes after parastomal hernia repairs in Denmark from 2007-2017 focusing on readmission and reoperation rates.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing parastomal hernia repair in Denmark from 2007-2017

Exclusion Criteria:

* If data is not fully registered in the Danish Hernia Database

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing parastomal hernia repair in Denmark from 2007-2017
Sampling Method: Non-Probability Sample
Enrollment: 1062 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Reoperation | 30 days
  Number of patients re-operated for a complication after a parastomal hernia repair

SECONDARY OUTCOMES:
Readmission | 90 days
  Number of patients readmitted after parastomal hernia repair
Recurrence | 10 years
  Number of patients operated for recurrence after a parastomal hernia repair

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Henriksen, Principal Investigator — Zealand University Hospital, Koege, Dept. of Surgery
Locations (1):
- Dept. of surgery, Køge Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No